CLINICAL TRIAL: NCT05000684
Title: A Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Initial Efficacy of Recombinant Humanized Anti-BTLA Monoclonal Antibody (JS004) Injection Combined With Toripalimab in Patients With Advanced Lung Cancer
Brief Title: Study of JS004 Combined With Toripalimab for Advanced Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS004-006-I/II-LC
Record Dates: First submitted 2021-08-10; First posted 2021-08-11 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Advanced Lung Cancer
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS004 200 mg in combination with toripalimab 240 mg was administered every 3 weeks as planned (Experimental)
  Interventions: Drug: JS004 in combination with toripalimab

INTERVENTIONS:
Drug: JS004 in combination with toripalimab — Usage and dosage: 200mg of JS004 combined with 240mg of JS001 is given every 3 weeks
  Other Names: JS004+JS001

SUMMARY:
This is an open-label phase I/II study to evaluate the safety, tolerability, pharmacokinetics and initial efficacy of JS004 injection combined with toripalimab in patients with advanced lung cancer who have failed standard therapy.

ELIGIBILITY:
Inclusion Criteria：

1. Sign the informed consent form voluntarily;
2. Age greater than or equal to 18 years old at time of signing informed consent, males and females are included;
3. Expected survival time is greater than or equal to 3 months;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
5. Pathologically confirmed locally advanced (Stage III B/C), metastatic or recurrent (Stage IV) non-small cell lung cancer (NSCLC);
6. Pathologically confirmed extensive-stage small cell lung cancer (ES-SCLC, according to the Veterans Administration Lung Study Group (VALG) staging system);
7. At least one measurable lesion as a target lesion (RECIST v1.1 criteria);
8. Agree to provide tumor tissue samples (provide fresh biopsy samples before treatment as far as possible，provide archived samples within 2 years for patients who cannot provide fresh biopsy samples before treatment;
9. The subject has good organ function as indicated by screening laboratory results；
10. Males of reproductive potential or females of childbearing potential must use effective contraceptive methods (such as oral contraceptives, intrauterine device or barrier method combined with spermicide) during the trial and continue contraception for 6 months after the end of treatment;
11. Good compliance and cooperated with the follow-up；

Exclusion Criteria:

1. Within 2 years prior to enrollment, had other active neoplasm malignancies except for the study disease, but excluding neoplasm malignancies expected to be cured after treatment (including but not limited to thyroid cancer, carcinoma cervix in situ, basal or squamous cell skin carcinoma, or ductal carcinoma in situ after radical surgery after adequate treatment);
2. Patients previously treated with anti-BTLA or anti-HVEM antibodies;
3. Patients previously discontinued treatment due to PD-1/PD-L1 inhibitor toxicity;
4. Adverse reaction caused by prior treatment that has not recovered to CTCAE Grade 1 and below (except Grade 2 toxicity that is long-lasting, not recoverable, and does not increase safety risk);
5. Received allogeneic hematopoietic stem cell transplantation or solid organ transplantation in the past;
6. A large amount of hydrothorax or ascites or pericardial effusion with clinical symptoms or requiring symptomatic treatment;
7. Known history of Lung disorder: history of Interstitial pneumonia/drug-induced interstitial Pneumopathy or pneumonia, symptomatic Bronchospasm;
8. Active infection requiring systemic therapy;
9. A positive result for human immunodeficiency virus (HIV) antibody test;
10. Known active tuberculosis (TB). For patients with suspicion of active TB should perform the test of chest X-ray, sputum, clinical signs and symptoms to exclude；
11. Have a history of psychotropic drug abuse and unable to withdraw or have mental disorders;
12. Pregnant or lactating woman;
13. Known to be allergic to JS004 or toripalimab and its components;
14. Other severe, acute or chronic medical or psychiatric disorders or laboratory abnormalities that, in the investigator's opinion, may increase the risk associated with study participation or may interfere with the interpretation of study results；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events (AE) and serious adverse events (SAE) were assessed | 2 years
  Incidence and severity of adverse events (AE) and serious adverse events (SAE) as assessed according to NCI-CTCAE 5.0, as well as abnormalities in vital signs, electrocardiogram, and laboratory tests

SECONDARY OUTCOMES:
OS | 2 years
  Duration of Response
DOR | 2 years
  Duration of Response
DCR | 2 years
  Disease Control Rate
PFS | 2 years
  Progression-free survival
Cmax | 2 years
  Maximum Plasma Concentration
Tmax | 2 years
  Time to Cmax
AUC0-t | 2 years
  Area under the concentration versus time curve from time 0 to the last measurable concentration
AUC0-inf | 2 years
  AUC from time 0 to infinity
Kel | 2 years
  Elimination rate constant
t1/2 | 2 years
  Elimination half life time
CL/F | 2 years
  Clearance
Vd/F | 2 years
  Apparent volume of distribution
Rac | 2 years
  Accumulation factor

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jilin Cancer Hospital, Changchun, Jilin
  - Cancer Hospital of Chinese Academy of Medical Sciences, Beijing